CLINICAL TRIAL: NCT03742063
Title: Clinical Evaluation of Neoadjuvant Chemotherapy for Primary Malignant Sarcomas That Originate in Bone: a Multi-center Retrospective Study for Standardization and Modification of Response Evaluation Criteria
Brief Title: Clinical Evaluation of Neoadjuvant Chemotherapy for Primary Malignant Sarcomas That Originate in Bone
Acronym: CESOFB-00
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CBTRA-00
Record Dates: First submitted 2018-11-11; First posted 2018-11-15 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Clinical Response; Histopathological Response; Prognosis
Keywords: osteosarcoma; Ewing sarcoma; clinical evaluation; pathological evaluation; chemotherapy; targeted therapy
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Huvos group I: Upon histopathological examination, the tumor response was assessed on the basis of the presence and extent of necrosis, which was assessed by a combination of gross and microscopic observations. Tumor necrosis was graded as per Picci et al. tumor histopathological response grading (Huvos classification), where grade I is 0% to 49%.
  Interventions: Drug: first-line chemotherapy
- Huvos group II: Upon histopathological examination, the tumor response was assessed on the basis of the presence and extent of necrosis, which was assessed by a combination of gross and microscopic observations. Tumor necrosis was graded as per Picci et al. tumor histopathological response grading (Huvos classification), where grade II is 50% to 89%.
  Interventions: Drug: first-line chemotherapy
- Huvos group III: Upon histopathological examination, the tumor response was assessed on the basis of the presence and extent of necrosis, which was assessed by a combination of gross and microscopic observations. Tumor necrosis was graded as per Picci et al. tumor histopathological response grading (Huvos classification), where grade III is 90% to 99%.
  Interventions: Drug: first-line chemotherapy
- Huvos group IV: Upon histopathological examination, the tumor response was assessed on the basis of the presence and extent of necrosis, which was assessed by a combination of gross and microscopic observations. Tumor necrosis was graded as per Picci et al. tumor histopathological response grading (Huvos classification), where grade IV is 100% necrosis.
  Interventions: Drug: first-line chemotherapy

INTERVENTIONS:
Drug: first-line chemotherapy — patients who routinely received neoadjuvant chemotherapy according to Peking University People's Hospital chemo-protocols (PKUPH-OS and PKUPH-ES)

SUMMARY:
For bone lesions treated with chemotherapy or targeted therapy, particularly for sarcomas that originate in bones, Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 is spurious because bone lesions are typically located in irregularly shaped bones, are difficult to measure accurately, and usually respond more slowly to treatment than soft tissue lesions. Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) allows for response to be measured in the absence of anatomic changes through assessment of metabolic activity. It does not, however, account for morphologic changes. This study evaluated whether clinical imaging findings of sarcomas after preoperative chemotherapy correlate with tumor responses by pathological evaluation using the rate of necrosis to develop reliable and quantitative clinical response criteria.

DETAILED DESCRIPTION:
We reviewed a total of 190 primary lesions by clinical imaging, including X-ray, computed tomography (CT), magnetic resonance imaging, and bone scan or PET/CT in patients who received neoadjuvant chemotherapy. All patients had curative surgery of those lesions at Peking University People's Hospital or Peking University Shougang Hospital. Pathological evaluation was completed by determination of the tumor necrosis rate following Huvos' description. We also performed statistical diversity analysis for different pathological groups and generated receiver operating characteristic curves (ROC) to define the thresholds to distinguish different pathological groups.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients with high-grade sarcoma that originated in bone and confirmed histologically;
* (2) patients who routinely received neoadjuvant chemotherapy according to Peking University People's Hospital chemo-protocols (PKUPH-OS and PKUPH-ES);
* (3) patients who had primary tumor resection with assessment of histological response according to literatures;
* (4) patients who had intact pre- and post-neoadjuvant chemotherapy imaging, which included X-ray, contrasted computed tomography (CT), and magnetic resonance imaging (MRI) of the primary lesions as well as chest CT (with each layer ≤5 mm), bone scan, or [18F]2-fluoro-2-deoxy-D-glucose-positron emission tomography (FDG-PET);
* (5) patients for whom follow-up information and evaluation after chemotherapy were available.

Exclusion Criteria:

* patients with incomplete medical materials;
* patients without surgery of the primary site/ without pathological analysis of the specimens;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively reviewed medical records of 190 patients with high-grade sarcomas (mainly osteosarcomas and Ewing's sarcomas) that originated in bone, who received neoadjuvant chemotherapy from June 1, 2014, to March 1, 2017, at Peking University People's Hospital and Peking University Shougang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Tumor necrosis rate | 2-3 months
  We evaluated all surgical resection specimens and were blinded to the clinical status. Upon histopathological examination, the tumor response was assessed on the basis of the presence and extent of necrosis, which was assessed by a combination of gross and microscopic observations. Tumor necrosis was graded as per Picci et al. tumor histopathological response grading (Huvos classification), where grade I is 0% to 49%, grade II is 50% to 89%, grade III is 90% to 99%, and grade IV is 100% necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Ph.D. and M.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moertel CG, Hanley JA. The effect of measuring error on the results of therapeutic trials in advanced cancer. Cancer. 1976 Jul;38(1):388-94. doi: 10.1002/1097-0142(197607)38:13.0.co;2-a. PMID 947531
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Choi H, Charnsangavej C, Faria SC, Macapinlac HA, Burgess MA, Patel SR, Chen LL, Podoloff DA, Benjamin RS. Correlation of computed tomography and positron emission tomography in patients with metastatic gastrointestinal stromal tumor treated at a single institution with imatinib mesylate: proposal of new computed tomography response criteria. J Clin Oncol. 2007 May 1;25(13):1753-9. doi: 10.1200/JCO.2006.07.3049. PMID 17470865
- [Background] Hamaoka T, Madewell JE, Podoloff DA, Hortobagyi GN, Ueno NT. Bone imaging in metastatic breast cancer. J Clin Oncol. 2004 Jul 15;22(14):2942-53. doi: 10.1200/JCO.2004.08.181. PMID 15254062
- [Background] Smith AD, Shah SN, Rini BI, Lieber ML, Remer EM. Morphology, Attenuation, Size, and Structure (MASS) criteria: assessing response and predicting clinical outcome in metastatic renal cell carcinoma on antiangiogenic targeted therapy. AJR Am J Roentgenol. 2010 Jun;194(6):1470-8. doi: 10.2214/AJR.09.3456. PMID 20489085
- [Background] Smith AD, Lieber ML, Shah SN. Assessing tumor response and detecting recurrence in metastatic renal cell carcinoma on targeted therapy: importance of size and attenuation on contrast-enhanced CT. AJR Am J Roentgenol. 2010 Jan;194(1):157-65. doi: 10.2214/AJR.09.2941. PMID 20028918
- [Background] Tsuchida Y, Therasse P. Response evaluation criteria in solid tumors (RECIST): new guidelines. Med Pediatr Oncol. 2001 Jul;37(1):1-3. doi: 10.1002/mpo.1154. No abstract available. PMID 11466715
- [Background] Costelloe CM, Chuang HH, Madewell JE, Ueno NT. Cancer Response Criteria and Bone Metastases: RECIST 1.1, MDA and PERCIST. J Cancer. 2010 Jun 28;1:80-92. doi: 10.7150/jca.1.80. PMID 20842228
- [Background] Bajpai J, Kumar R, Sreenivas V, Sharma MC, Khan SA, Rastogi S, Malhotra A, Gamnagatti S, Kumar R, Safaya R, Bakhshi S. Prediction of chemotherapy response by PET-CT in osteosarcoma: correlation with histologic necrosis. J Pediatr Hematol Oncol. 2011 Oct;33(7):e271-8. doi: 10.1097/MPH.0b013e31820ff78e. PMID 22193290
- [Background] Byun BH, Kim SH, Lim SM, Lim I, Kong CB, Song WS, Cho WH, Jeon DG, Lee SY, Koh JS, Chung SK. Prediction of response to neoadjuvant chemotherapy in osteosarcoma using dual-phase (18)F-FDG PET/CT. Eur Radiol. 2015 Jul;25(7):2015-24. doi: 10.1007/s00330-015-3609-3. Epub 2015 Feb 14. PMID 25680716
- [Background] Bajpai J, Gamnagatti S, Kumar R, Sreenivas V, Sharma MC, Khan SA, Rastogi S, Malhotra A, Safaya R, Bakhshi S. Role of MRI in osteosarcoma for evaluation and prediction of chemotherapy response: correlation with histological necrosis. Pediatr Radiol. 2011 Apr;41(4):441-50. doi: 10.1007/s00247-010-1876-3. Epub 2010 Oct 27. PMID 20978754
- [Background] Lamuraglia M, Raslan S, Elaidi R, Oudard S, Escudier B, Slimane K, Penna RR, Wagner M, Lucidarme O. mTOR-inhibitor treatment of metastatic renal cell carcinoma: contribution of Choi and modified Choi criteria assessed in 2D or 3D to evaluate tumor response. Eur Radiol. 2016 Jan;26(1):278-85. doi: 10.1007/s00330-015-3828-7. Epub 2015 May 8. PMID 25953002
- [Background] O JH, Lodge MA, Wahl RL. Practical PERCIST: A Simplified Guide to PET Response Criteria in Solid Tumors 1.0. Radiology. 2016 Aug;280(2):576-84. doi: 10.1148/radiol.2016142043. Epub 2016 Feb 24. PMID 26909647
- [Background] Rosen G, Caparros B, Huvos AG, Kosloff C, Nirenberg A, Cacavio A, Marcove RC, Lane JM, Mehta B, Urban C. Preoperative chemotherapy for osteogenic sarcoma: selection of postoperative adjuvant chemotherapy based on the response of the primary tumor to preoperative chemotherapy. Cancer. 1982 Mar 15;49(6):1221-30. doi: 10.1002/1097-0142(19820315)49:63.0.co;2-e. PMID 6174200